CLINICAL TRIAL: NCT04466943
Title: The Impact of Moderate Versus Deep Neuromuscular Blockade on Enhanced Recovery After Bariatric Anesthesia: A Randomized Double Blinded Clinical Trial
Brief Title: The Impact of Moderate Versus Deep Neuromuscular Blockade on Enhanced Recovery After Bariatric Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Narjes Sultan AL-Otaibi, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: E-19-3960
Record Dates: First submitted 2020-06-29; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the attending anesthesiologist and anesthesia assistant are going to be aware of the allocation in order to administer the required level of NMB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): Moderate neuromuscular blockade (NMB) , defined as a 1±2 twitch response to the train-of four (TOF) by stimulation of the ulnar nerve. The device which will be used is neuromuscular transmission monitor (NMT) to test the depth of muscle relaxation after giving rocuronium which is a muscle relaxant during general anesthesia.
  Interventions: Device: Neuromuscular transmission monitoring (NMT)
- group B (Experimental): Deep NMB, defined by (0 twitch count in the TOF, 1±2 twitch responses in the post-tetanic count. The device which will be used is neuromuscular transmission monitor (NMT) to test the depth of muscle relaxation after giving rocuronium which is a muscle relaxant during general anesthesia.
  Interventions: Device: Neuromuscular transmission monitoring (NMT)

INTERVENTIONS:
Device: Neuromuscular transmission monitoring (NMT) — NMT is to monitor the depth of neuromuscular blockade intensity
  Other Names: NMT monitor the depth of muscle relaxation and based upon its reading Rocuronium which is muscle relaxant to be given to the patient under general anesthesia

SUMMARY:
Most published articles suggest that deep neuromuscular blockade is required for bariatric surgery. However, the evidence for such practice is still inconclusive. From the clinical experience at a major bariatric center of volume exceeding six hundred procedures annually, the investigators believe that moderate neuromuscular blockade will provide an adequate surgical condition and significantly facilitate enhanced recovery after bariatric procedures.

DETAILED DESCRIPTION:
Muscle relaxation is paramount for successful laparoscopic surgery. However the optimal degree of neuromuscular blockade (NMB) is not identified yet. Previous studies showed conflicting results on the outcomes of laparoscopic surgical conditions when moderate NMB was compared to deep blockade .The evidence for the use of either modalities is rather limited . In the recent literature, there is insufficient evidence to conclude that deep NMB improves surgical conditions during laparoscopic bariatric surgery.

In the recent literature, there is insufficient evidence to conclude that deep NMB improves surgical conditions during laparoscopic bariatric surgery. However postoperative pulmonary function was decreased independently of the depth of NMB regime. There are limited data on the effect of such practices on postoperative outcomes especially in enhanced recovery after bariatric anesthesia (ERABA) .A previous study by Unterbuchner C has showed deep NMB may improve surgical conditions during low-pressure capnoperitoneium , However ,it has also been reported by M.H. Bruintjes and his colleagues showed that the routine capnoperitoneium insufflation pressure improved surgical conditions independent of the level of muscular relaxation. Torensma B and his colleagues have reported that the previous pregnancy can affects the abdominal wall strength and eventually the degree of relaxation Therefore, the investigators have decided to exclude any females with previous history of pregnancy in the study design and also report interaction between inhalation anesthetics and NMB, through augmentation of the effect of NMB.

Martini and his colleagues showed that , rating of the quality of surgical conditions considerably varies between different surgeons when assessed through Leiden-Surgical-Rating-scale . Therefor in this study, the Lieden-surgical-score is going to be used by the bariatric surgeon who is going to be the operating consultant in this study population.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years.
2. Obese or morbidly obese as defined by a BMI > 35 (kg/m2).
3. American Society of Anesthesiologists physical status class II, or III.
4. Presenting of Laparoscopic sleeve gastrectomy.

Exclusion Criteria:

1. History of allergy to Rocuronium or Sugammadex.
2. History of allergy to Dexamethasone, Ondansetron, Paracetamol, Fentanyl, Propofol, Morphine or Tramadol.
3. Current or previous pregnancy.
4. History of renal impairment, (We are going to use the Cockcroft-Gault equation is the gold standard for estimating renal function for the purposes of drug dosing cut off point: CrCl/GFR=30ml/min) The GFR calculator is available at: http://clincalc.com/Kinetics/CrCl.aspx?example
5. Patient on oxygen therapy , e,g CPAP

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete recovery in post anesthesia care unit (PACU) without residual curarization | immediate postoperative in the PACU
  clinical signs of recovery are met in the PACU

SECONDARY OUTCOMES:
Complete recovery in the ward | first postoperative day
  clinical signs of recovery are met in the ward

CONTACTS AND LOCATIONS:
Overall Officials: ALHARBI, Principal Investigator — KindSaudU
Locations (1):
- King Saud University College of Medicine and King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
to be submit
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: i year
Access Criteria: to be submit